CLINICAL TRIAL: NCT03095677
Title: Acute and Chronic Effects of Dynamic Apnea in Healthy Untrained Subjects
Acronym: APNEX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Régional d'Orléans (Other)
Collaborators: Laboratoire de Complexité, Innovation et Activités Motrices et Sportives (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: CHRO-2015-01
Record Dates: First submitted 2016-09-27; First posted 2017-03-30 (Actual); Last update posted 2018-05-07 (Actual); Status verified 2018-05

CONDITIONS: Apnea
Keywords: dynamic apnea; muscle oxygenation; physical performance
MeSH Terms: conditions — Apnea | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Apnea Group (GApn) (Experimental): Program of training with exercises including apneas
  Interventions: Other: Program of training with exercises including apnea
- Control Group (GC) (Other): Program of training with exercises without apnea
  Interventions: Other: Program of training with exercises without apnea

INTERVENTIONS:
Other: Program of training with exercises including apnea — 16 training session on cycle ergometry with exercises including apneas.
  Arms: Apnea Group (GApn)
Other: Program of training with exercises without apnea — 16 training session on cycle ergometry with exercises without apnea
  Arms: Control Group (GC)

SUMMARY:
The inclusion of short periods of apnea (several seconds) during exercise (i.e. dynamic apnea) induces a significant decrease in blood oxygenation and muscle tissue. To date, the immediate effects ("acute apnea") of this decrease in the quantity of oxygen available at the muscle and brain level are poorly understood. Moreover, a physical training during which these short periods of apnea ("chronic apnea") would be included could lead to physiological adaptations and to improvement in physical performance similar to those obtained during altitude training.

The purpose of this study is to evaluate the effects of acute dynamic apnea on metabolism.

ELIGIBILITY:
Inclusion Criteria:

* The cutaneous thickness at the vastus lateralis level lower than 1.5 cm to obtain the reliable muscle oxygenation measurement
* Subjects will have to sign the inform consent before the beginning of the study

Exclusion Criteria:

* Contraindications to regular physical exercise practice
* To practice an endurance sport more than 1h/week
* Regular practice of apnea
* Chronic use of cannabis and/or alcohol
* Cardiac or metabolic pathology
* Asthma and/or bronchodilatator treatment
* ECG abnormality at rest
* Regular consumption of tobacco

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2016-04-08 (Actual); Primary Completion 2017-11-20 (Actual); Study Completion 2017-11-20 (Actual)

PRIMARY OUTCOMES:
Spectometry to measure hemoglobin rate | 3 weeks
  Measurement of oxygenation
Wingate test to measure maximum consumption of dioxygen | 3 weeks
  Measurement of aerobic performance
Measurement of hormonal markers | 3 weeks
  Measurement of Dehydroepiandrostenedione (DHEA)
Jaeger debimeter system to measure of peak oxygen | 3 weeks
  Measurement of oxygen consumptiom
Measurement of arterial saturation in dioxygen | 3 weeks
  Measurement by ear blood micro-sample
Spectometry to measure hemoglobin | 12 weeks
  Measurement of oxygenation
Measurement of hormonal markers | 12 weeks
  Measurement of Dehydroepiandrostenedione (DHEA)
Jaeger debimeter system to measure of peak oxygen | 12 weeks
  Measurement of oxygen consumption,
Measurement of arterial saturation in dioxygen | 12 weeks
  Measurement by ear blood micro-sample

SECONDARY OUTCOMES:
Cardiac frequency | 3 weeks
  measurement with a 12 lead - Electrocardiogamm
Cardiac frequency | 12 weeks
  measurement with a 12 lead - Electrocardiogramm
Borg scale to measure penibility of the effort | week 3
Borg scale to measure penibility of the effort | week 12

CONTACTS AND LOCATIONS:
Overall Officials: Virgile AMIOT, Ph, Principal Investigator — CHR ORLEANS
Locations (1):
- CHR d'Orléans, Orléans, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Andersson JP, Liner MH, Runow E, Schagatay EK. Diving response and arterial oxygen saturation during apnea and exercise in breath-hold divers. J Appl Physiol (1985). 2002 Sep;93(3):882-6. doi: 10.1152/japplphysiol.00863.2001. PMID 12183481
- [Background] Caquelard F, Burnet H, Tagliarini F, Cauchy E, Richalet JP, Jammes Y. Effects of prolonged hypobaric hypoxia on human skeletal muscle function and electromyographic events. Clin Sci (Lond). 2000 Mar;98(3):329-37. PMID 10677392
- [Background] de Bruijn R, Richardson M, Schagatay E. Increased erythropoietin concentration after repeated apneas in humans. Eur J Appl Physiol. 2008 Mar;102(5):609-13. doi: 10.1007/s00421-007-0639-9. Epub 2007 Dec 19. PMID 18097682
- [Background] Dufour SP, Ponsot E, Zoll J, Doutreleau S, Lonsdorfer-Wolf E, Geny B, Lampert E, Fluck M, Hoppeler H, Billat V, Mettauer B, Richard R, Lonsdorfer J. Exercise training in normobaric hypoxia in endurance runners. I. Improvement in aerobic performance capacity. J Appl Physiol (1985). 2006 Apr;100(4):1238-48. doi: 10.1152/japplphysiol.00742.2005. PMID 16540709